CLINICAL TRIAL: NCT03050710
Title: A Prospective, Open-label, Multicenter, Post-market Study Evaluating Princess® VOLUME Lidocaine for the Correction of Nasolabial Folds
Brief Title: Princess® VOLUME Lidocaine for the Correction of Nasolabial Folds
Acronym: VINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPH-401-201258
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2018-08

CONDITIONS: Nasolabial Fold, Hypoplastic

STUDY DESIGN:
Intervention Model Description: Princess® VOLUME Lidocaine for the correction of nasolabial folds
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Princess® VOLUME Lidocaine (Other): Princess® VOLUME Lidocaine is administered by injection into the deep dermis or subcutis. The volume applied depends on the size of the area which requires correction and will be selected by the investigator, but will not exceed 10 mL in total per treatment. A single application, with optional Touch-up treatment after two weeks, if the desired level of correction has not been achieved with the initial applicatio
  Interventions: Device: Princess® VOLUME Lidocaine

INTERVENTIONS:
Device: Princess® VOLUME Lidocaine — Princess® VOLUME Lidocaine injections up to 10 ml given to the patients at baseline, and touch-up at week 2, if applicable

SUMMARY:
In this study, eligible subjects with moderate to severe nasolabial folds will be treated with Princess® VOLUME Lidocaine and will return for follow-up assessments 2, 4, 24 and 36 weeks after the treatment. A Touch-up treatment may be done at Week 2, if deemed appropriate by the investigator.

DETAILED DESCRIPTION:
This is a prospective, open label, multicenter, post-market investigation. Following informed consent and screening, eligible subjects with moderate to severe nasolabial folds will be treated with Princess® VOLUME Lidocaine, and will return for follow-up assessments 2, 4, 24 and 36 weeks after the treatment. A Touch-up treatment may be done at Week 2, if deemed appropriate by the investigator. The performance of the investigational device will be evaluated by the investigator by assessing severity of nasolabial folds using the Nasolabial Folds Severity Rating Scale (NLF-SRS) (4, 24 and 36 weeks after the treatment and in comparison to Day 0), global aesthetic improvement (4, 24 and 36 weeks after the treatment). The subject will evaluate pain intensity associated with the treatment (at Day 0 and at Week 2 (if Touch-up treatment occurred)), and satisfaction with the treatment 4, 24 and 36 weeks after the treatment.

The safety will be evaluated based on occurrence of adverse events, which will be collected throughout the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older
2. Presence of two fully visible, approximately symmetrical nasolabial folds, with each of the folds scored 2-3 according to the 5-grade Nasolabial Folds Severity Rating Scale (NLF-SRS) as assessed by the investigator
3. Healthy skin in the facial area and free of diseases that could interfere in cutaneous aging evaluation
4. Willingness to abstain from any aesthetic or surgical procedures in the treatment area for the duration of the clinical investigation
5. Written signed and dated informed consent

Exclusion Criteria:

1. Pregnancy, lactation, planned pregnancy or unwillingness to use contraception at any time during the study (for women of child-bearing potential only)
2. History of mental disorders or emotional instability
3. History of allergic reaction or hypersensitivity to hyaluronic acid, lidocaine, or any amide-based anaesthetic
4. Presence of silicone implant or another non-absorbable substance (permanent fillers) in the nasolabial region
5. Facial surgery or implantation of dermal fillers, absorbable and nonabsorbable sutures (thread), laser therapy, dermoabrasion, or botulinum toxin application in the nasolabial region within previous 12 months, or chemical peeling within previous 3 months, or planning to undergo such procedures in the treatment area during the study
6. Presence of infectious, inflammatory, or proliferative lesions in the nasolabial region
7. Cutaneous lesions in the treatment area
8. Known human immune deficiency virus-positive individuals
9. History of allergies against aesthetic filling products and recurrent herpes simplex
10. Tendency to hypertrophic scars and/or keloid formation
11. History or presence of any autoimmune or connective tissue disease, or current treatment with immune therapy
12. Diabetes mellitus or uncontrolled systemic diseases
13. Use of anticoagulant, antiplatelet or thrombolytic medication from 10 days pre- to 3 days post injection
14. Any medical condition which, in the investigator's opinion. prohibits the inclusion in the study
15. Current or previous (within 30 days of enrolment) treatment with another investigational drug and/or medical device or participation in another clinical study
16. Previous enrolment in this clinical investigation
17. Subjects whose participation in clinical trials is prohibited by the Austrian Medical Devices Act (e.g., persons with a legal custodian appointed due to mental disability, prisoners, soldiers and other members of the armed forces, civil servants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medical University Graz, Graz
  - MÄZ WIEN Medizinisch Ästhetisches Zentrum Wien, Vienna
  - Ordination Dr. Rudolf Bartsch und Dr. Katrin Bartsch, Vienna

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 subjects were screened and enrolled.
Period: Overall Study
Arm/Group | Princess® VOLUME Lidocaine
Started | 62
Completed | 61
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 62 screened subjects were treated at least once with the investigational medical device and were included in the SAF.
  62 subjects had at least one post-treatment assessment and at least one NLF severity assessment based on the NLF-SRS and were included in the ITT population.
  One subject terminated the investigation early after Week 4 due to a clinical investigation plan (CIP) deviation.
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 62
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 62

OUTCOME MEASURES:

1. Primary Outcome: NLF-SRS Grade of Nasolabial Folds Change
Description: The average change versus baseline in the NLF-SRS grade of nasolabial folds at Week 24 as evaluated by the investigator.
  The Croma NLF-SRS is a validated, 5-point scale ranging from Grade 0 (none or minimal) to Grade 4 (extreme), therefore a reduction in value, represents an improvement on an aesthetical perspective
Time Frame: 24 weeks
Population: ITT - Intent to treat Population - as defined in Baseline Analysis Population Description
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 61
score on a scale | -1.50 (0.58)

2. Primary Outcome: NLF-SRS Grade of Nasolabial Folds Reduction
Description: The proportion of subjects with the NLF-SRS grade reduced by ≥1 point at week 24 versus baseline.
  The Croma NLF-SRS is a validated, 5-point scale ranging from Grade 0 (none or minimal) to Grade 4 (extreme), therefore a reduction in value, represents an improvement on an aesthetical perspective
Time Frame: 24 weeks
Population: ITT - Intent to treat Population - as defined in Baseline Analysis Population Description
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 61
Participants | 58

3. Secondary Outcome: NLF-SRS Grade of Nasolabial Folds Change - Other Timepoints
Description: The average change versus baseline in the NLF-SRS grade of nasolabial folds at Week 4 and Week 36 as evaluated by the investigator.
  The Croma NLF-SRS is a validated, 5-point scale ranging from Grade 0 (none or minimal) to Grade 4 (extreme), therefore a reduction in value, represents an improvement on an aesthetical perspective
Time Frame: Week 4, Week 36
Population: ITT - Intent to treat Population - as defined in Baseline Analysis Population Description
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
score on a scale
  Week 4: number analyzed (Participants) | 61
  Week 4 | -1.54 (0.62)
  Week 36 | -1.35 (0.66)

4. Secondary Outcome: NLF-SRS Grade of Nasolabial Folds Reduction- Other Timepoints
Description: The proportion of subjects with the NLF-SRS grade reduced by ≥1 point at week 4 and week 36 versus baseline
Time Frame: week 4, week 36
Population: ITT - Intent to treat Population - as defined in Baseline Analysis Population Description
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
Participants
  Week 4: number analyzed (Participants) | 61
  Week 4 | 58
  Week 36 | 54

5. Secondary Outcome: Aesthetic Improvement
Description: The proportion of subjects with aesthetic improvement at Week 4, Week 24 and Week 36, as evaluated by the investigator using the Global Aesthetic Improvement Scale (GAIS)
Time Frame: week 4, week 24, week 36
Population: ITT - Intent to treat Population - as defined in Baseline Analysis Population Description
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
Participants
  Week 4: number analyzed (Participants) | 61
  Week 4 | 61
  Week 24: number analyzed (Participants) | 61
  Week 24 | 58
  Week 36 | 58

6. Secondary Outcome: Subjects' Satisfaction With Aesthetic Outcome
Description: Subjects' satisfaction rate with aesthetic outcome of the treatment at Week 4, Week 24 and Week 36, as evaluated by the subject
Time Frame: week 4, week 24, week 36
Population: ITT - Intend to Treat Population as defined in the Baseline Analysis Population description. The results below reflect the subjects who rated their satisfaction with the treatment as 'very satisfied'.
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
Participants
  Week 4: number analyzed (Participants) | 61
  Week 4 | 52
  Week 24: number analyzed (Participants) | 61
  Week 24 | 48
  Week 36 | 49

7. Secondary Outcome: Pain Intensity
Description: The average pain intensity during and after the treatment, as evaluated by the subject using an 11-point numeric pain rating scale (NPRS), where 0= no pain and 10 = worst pain imaginable, immediately after the last injection and 15 minutes thereafter. Lower scores represent better outcomes (less pain). Higher scores represent worse outcomes (more pain).
Time Frame: Day 1, Day 15
Population: ITT - Intent to treat Population - defined in Baseline Analysis Population Description
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
score on a scale
  Baseline- Initial Assessment (right after injection) | 1.2 (1.3)
  Baseline - Second Assessment ( 15 min after injection) | 0.1 (0.4)
  Baseline - Change from initial assessment to second assessment | -1.0 (1.1)
  Week 2 /Touch up - Initial Assessment (right after injection): number analyzed (Participants) | 8
  Week 2 /Touch up - Initial Assessment (right after injection) | 1.5 (0.9)
  Week 2 /Touch up - Second Assessment ( 15 min after injection): number analyzed (Participants) | 8
  Week 2 /Touch up - Second Assessment ( 15 min after injection) | 0.0 (0.0)
  Week 2/ touch up - Change from initial assessment to second assessment: number analyzed (Participants) | 8
  Week 2/ touch up - Change from initial assessment to second assessment | -1.5 (0.9)

8. Secondary Outcome: NLF-SRS Grade of Nasolabial Folds Reduction- Imaging Independent Reviewer
Description: The proportion of subjects with the NLF-SRS grade reduced by ≥1 point versus Baseline at Week 24 as evaluated by the independent reviewer of photographs.
Time Frame: Week 24
Population: ITT- Intent to treat population - As defined in the Baseline Analysis Population Description
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 61
Participants | 60

9. Other Pre Specified Outcome: Safety Events
Description: Occurrence and frequency of adverse events
Time Frame: From day 0 until patient last visit / week 36
Population: SAF - as defined in the Baseline Analysis Population Description
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME Lidocaine
Number analyzed (Participants) | 62
Participants
  Adverse Device Effect - Injection site hematoma | 1
  Adverse Device Effect - Injection site hypoesthesia | 6
  Adverse Device Effect - Injection site pain | 2
  Adverse Device Effect - Syncope | 1
  Influenza | 1
  Lice Infestation | 1
  Rhinitis | 1
  Urinary tract infection | 1
  Ligament sprain | 1
  Synovitis | 1
  Polyneuropathy | 1

ADVERSE EVENTS:
Time Frame: 36 weeks - Up to 36 weeks after treatment (Day 0)
Description: AEs will be detected at each visit by clinical examination and by asking the subject about the occurrence of AEs. Care should be taken not to introduce bias when eliciting AE information from the subject. In addition, the subjects will be instructed to immediately contact the investigator/study site in case of occurrence of any untoward event between visits.
Arm/Group | Princess® VOLUME Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 12/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Princess® VOLUME Lidocaine (N=62)
injection site hypoaesthesia (General disorders) | 6 (6)
Injection site pain (General disorders) | 2 (2)
Injection site haematoma (General disorders) | 1 (1)
pyrexia (General disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
influenza (Infections and infestations) | 1 (1)
lice infestation (Infections and infestations) | 1 (1)
rhinitis (Infections and infestations) | 1 (1)
ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
polyneuropathy (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT03050710/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT03050710/SAP_001.pdf